CLINICAL TRIAL: NCT05197764
Title: The Integration of Macroscopic and Microscopic Muscle Properties With Cell Modelling to Feature Altered Neuromuscular Behavior in Cerebral Palsy: 3D-Macroscopic Muscle Architecture in Cerebral Palsy
Brief Title: Evaluation of Macroscopic Muscle Growth in Infants and Young Children With Spastic Cerebral Palsy
Acronym: 3D-MMAP
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Pulderbos revalidatiecentrum (Unknown); Revalidatieziekenhuis Inkendaal (Unknown)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62187
Record Dates: First submitted 2021-08-18; First posted 2022-01-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Spastic Cerebral Palsy; Acquired Brain Injury
Keywords: Spastic Cerebral Palsy; Acquired Brain Injury; Brain imaging; 3D freehand ultrasound; Muscle morphology; Range of motion; Stiffness; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with spastic cerebral palsy: Children between 6 months and 9 years old.
- Typically developing children: Children between 6 months and 9 years old.
- Children with an acquired brain injury: Children between 1,5 years and 9 years.

SUMMARY:
A mixed longitudinal design study will be carried out to explore the onset and time course of morphological muscle changes on a macroscopic level in children with spastic cerebral palsy (SCP). Therefore, this project aims to (1) describe the macroscopic morphological muscle changes with increasing age and (2) evaluate the onset and development of muscle alterations in relation to the brain lesion (e.g., timing, extent and location), to the neuromuscular impairments and to treatment. Overall, this project will evaluate the macroscopic muscle properties by means of 3D freehand ultrasound (3DfUS).

DETAILED DESCRIPTION:
Background:

Recent literature reviews have emphasized the need for longitudinal studies with multiple measurement time- points to properly identify the natural course of muscle growth in young children with SCP, compared to typically developing (TD) children. The etiology of SCP, including the underlying brain lesion, may also be relevant to understand the onset and early development of altered muscle growth. Since the perinatal brain lesion in congenital SCP results in early abnormal neuronal input to the muscle, the process of muscle formation and maturation is likely to be disturbed. Because the overall treatment goal is to improve and maintain the functional abilities of children with SCP, there is a growing interest in the relation between the brain lesions (defined by MRI) and motor outcomes. However, no studies have systematically explored the relation between intrinsic muscle alterations and the brain lesion characteristics.

Improved understanding of morphologically muscle changes during growth, and how the participants relate to the timing of the brain lesion, to clinical neuromuscular impairments and to treatment, has potential to classify SCP muscles into sub-groups, or phenotypes. Moreover, these insights can reveal new markers to optimize treatment protocols or develop new treatments, leading to patient-tailored treatment management and new avenues for improving function in children with SCP.

Aim:

The focus of this study is to improve insights in the onset, development and progression of morphological macroscopic muscle changes for growing children with spastic cerebral palsy. The diversity in macroscopic muscle growth will thereby be considered in longitudinal studies, starting shortly after the occurrence of the brain injury.

To achieve this general research goal, this project plans two main studies. In study 1, the aim is to evaluate macroscopic morphological muscle changes with age. In study 2, the aim is to evaluate these muscle alterations in relation to the brain lesion characteristics.

The first study is focused on longitudinal evaluation of macroscopic muscle properties with age. This project generally aim to define changes in muscle properties over 2 years of time in children with SCP of different age-groups and to compare the differences between children with SCP and TD children in these specific age-groups. This project hypothesizes that the development of macroscopic muscle properties is significantly altered between CP age-groups and between CP and TD children. As a sub-goal of the first study, this project will describe the rate of muscle specific changes in SCP (for two lower limb muscles), the differences in rate of changes between three GFMCS levels and the impact of the number of previous Botulinum neurotoxin A (BoNT-A) injections on the rate of changes.

The second study is focused on the longitudinal muscle changes started from the early years of life. This altered muscle growth will be related to the brain lesion characteristics (i.e., timing, extent and location). This project hypothesizes that the onset and progress of these muscle changes is different between patient groups, which are defined by the age of the patients at the event of the brain lesion. With the majority of SCP brain lesions occurring during the last trimester of pregnancy, it can be hypothesized that the early timing of brain lesion and thus an early abnormal neuronal input to the muscle influences muscle development, suggesting a primary nature of altered muscle growth.

The main outcome of this research project is the evaluation of muscle changes in children with brain lesion. The primary muscle parameters are muscle volume, muscle belly length and echo-intensity of two lower limb muscles.

Methods/design:

Study 1: Children will enter at different ages, ranging from 2 till 9 years of age, and will participate in a 2-years follow-up with one year time interval. The children with SCP will be equally distributed between age-groups (2-5 and 6-9 years). Only children with a gross motor function level of one, two or three will be included. For this study, 80 children with congenital CP and 60 aged-matched TD children will be included.

Study 2: Two patient groups of children will be included (1) children with congenital CP (aged between 6 months and 3 years) with a brain lesion that occurred before or around birth and (2) children with acquired brain injury (ABI) (aged between 1,5 and 9 years), with a brain lesion that occurred at least one year after birth. All children will be enrolled at least 6 months after the occurrence of the brain injury and will be assessed over a 2-year period with 5 measurement time points (every 6 months). This project aims to include 48 children with congenital CP, 16 children with ABI and 25 TD children.

Participants will be evaluated at the University Hospitals Leuven (UZ Leuven) at campus Gasthuisberg or campus Pellenberg and the rehabilitation centers of Pulderbos and Inkendaal. Data will be collected during a hospital visit and every participant will undergo at least a 3DfUS measurement of the medial gastrocnemius and the semitendinosus muscle. Other information that will be collected out of the available medical records includes the results of the structural brain MRI, the use of medication, treatment details (physiotherapy, orthotics and/or orthopedic interventions), anthropometric measures (body weight and length and leg lengths), data of a standard clinical examination (joint range of motion, spasticity, muscle selectivity and strength), data of a neurological examination more specific the Hammersmith Infant Neurological Examination (HINE) and the motor development by using the Motor Scales of the Bayley-III-NL.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of spastic cerebral palsy or patients at high-risk for spastic cerebral palsy
* Suspected GMFCS levels I-III (GMFCS = Gross Motor Function Classification Scale, expressing the overall functional level of impairment)

Exclusion Criteria:

* Non-ambulatory
* Botulinum neurotoxin type-A injections six months prior to enrollment
* Lower limb surgery two years prior to enrollment
* Muscle surgery at the muscles in the lower limb
* Selective dorsal rhizotomy as treatment history
* Presence of ataxia or dystonia
* Severe co-morbidities (severe epilepsy, severe behavior problems that impede the cooperation)

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with spastic cerebral palsy, who have routine follow-up care at the CP reference center of the University Hospitals Leuven, the rehabilitation centers of Pulderbos and/or Inkendaal
Sampling Method: Non-Probability Sample
Enrollment: 229 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall change in muscle volume of the medial gastrocnemius muscle and the semitendinosus muscle | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Estimation of the muscle belly volume by 3DfUS. Muscle volume will be normalized to anthropometric growth.
Overall change in muscle length of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Estimation of the muscle belly length, tendon length and muscle tendon unit complex length by 3DfUS. Muscle lengths will be normalized to anthropometric growth.
Overall change in muscle echo-intensity of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Estimation of the echo-intensity by 3DfUS.
Evaluation of the brain lesion based on MRI imaging | Once during the study participation of 2 years.
  Estimation of the type, extend and location of the brain lesion by MRI imaging assessment tool (Fiori scale)

SECONDARY OUTCOMES:
Overall change of range of motion of the ankle and knee joint | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Evaluation by goniometry
Overall change of spasticity of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Evaluation by Modified Ashworth Scale. This scale has a score from 0 to 4. If the score is higher, the muscle has more spasticity.
Overall change of muscle strength of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Evaluation by manual muscle testing with a score from 0 to 5. If the score is higher, the muscle is stronger.
Overall change of muscle selectivity of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Evaluation by Selective Control Assessment of the Lower Extremity (SCALE) clinical tool. This scale has a score from 0 to 2. If the score is higher, the muscle selectivity is better.
Physiotherapy | Through a study participation of 2 years, with an evaluation moment every 6 months.
  The frequency, duration and content of the physiotherapy sessions that the patients receive as their standard of care will be taken into account for the interpretation of the results.
Orthotics | Through a study participation of 2 years, with an evaluation moment every 6 months.
  The type, frequency and duration of the orthotics' use, both during day and night will be taken into account for the interpretation of the results
Change in fascicle length of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Estimation of the fascicle length by 2D and 3DfUS
Overall change in pennation angle of the medial gastrocnemius muscle and the semitendinosus muscle. | Through a study participation of 2 years, with an evaluation moment every 6 months.
  Estimation of the pennation angle by 2D and 3DfUS.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Prof. dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mockford M, Caulton JM. The pathophysiological basis of weakness in children with cerebral palsy. Pediatr Phys Ther. 2010 Summer;22(2):222-33. doi: 10.1097/PEP.0b013e3181dbaf96. PMID 20473109
- [Background] Theis N, Mohagheghi AA, Korff T. Mechanical and material properties of the plantarflexor muscles and Achilles tendon in children with spastic cerebral palsy and typically developing children. J Biomech. 2016 Sep 6;49(13):3004-3008. doi: 10.1016/j.jbiomech.2016.07.020. Epub 2016 Jul 26. PMID 27515440
- [Background] Gough M, Shortland AP. Could muscle deformity in children with spastic cerebral palsy be related to an impairment of muscle growth and altered adaptation? Dev Med Child Neurol. 2012 Jun;54(6):495-9. doi: 10.1111/j.1469-8749.2012.04229.x. Epub 2012 Feb 27. PMID 22364585
- [Background] Mathewson MA, Lieber RL. Pathophysiology of muscle contractures in cerebral palsy. Phys Med Rehabil Clin N Am. 2015 Feb;26(1):57-67. doi: 10.1016/j.pmr.2014.09.005. PMID 25479779
- [Background] Sarnat HB. Cerebral dysgeneses and their influence on fetal muscle development. Brain Dev. 1986;8(5):495-9. doi: 10.1016/s0387-7604(86)80093-6. PMID 3541664
- [Background] Baldwin KM, Haddad F. Effects of different activity and inactivity paradigms on myosin heavy chain gene expression in striated muscle. J Appl Physiol (1985). 2001 Jan;90(1):345-57. doi: 10.1152/jappl.2001.90.1.345. PMID 11133928
- [Background] Cenni F, Schless SH, Bar-On L, Aertbelien E, Bruyninckx H, Hanssen B, Desloovere K. Reliability of a clinical 3D freehand ultrasound technique: Analyses on healthy and pathological muscles. Comput Methods Programs Biomed. 2018 Mar;156:97-103. doi: 10.1016/j.cmpb.2017.12.023. Epub 2017 Dec 22. PMID 29428080
- [Background] Haberfehlner H, Maas H, Harlaar J, Becher JG, Buizer AI, Jaspers RT. Freehand three-dimensional ultrasound to assess semitendinosus muscle morphology. J Anat. 2016 Oct;229(4):591-9. doi: 10.1111/joa.12501. Epub 2016 Jun 6. PMID 27271461
- [Result] De Beukelaer N, Vandekerckhove I, Molenberghs G, Naulaers G, Thewissen L, Costamagna D, Van Campenhout A, Desloovere K, Ortibus E. Longitudinal trajectory of medial gastrocnemius muscle growth in the first years of life. Dev Med Child Neurol. 2024 Apr;66(4):531-540. doi: 10.1111/dmcn.15763. Epub 2023 Oct 3. PMID 37786988
- [Result] De Beukelaer N, Vandekerckhove I, Huyghe E, Molenberghs G, Peeters N, Hanssen B, Ortibus E, Van Campenhout A, Desloovere K. Morphological Medial Gastrocnemius Muscle Growth in Ambulant Children with Spastic Cerebral Palsy: A Prospective Longitudinal Study. J Clin Med. 2023 Feb 16;12(4):1564. doi: 10.3390/jcm12041564. PMID 36836099
- [Result] De Beukelaer N, Weide G, Huyghe E, Vandekerckhove I, Hanssen B, Peeters N, Uytterhoeven J, Deschrevel J, Maes K, Corvelyn M, Costamagna D, Gayan-Ramirez G, Van Campenhout A, Desloovere K. Reduced Cross-Sectional Muscle Growth Six Months after Botulinum Toxin Type-A Injection in Children with Spastic Cerebral Palsy. Toxins (Basel). 2022 Feb 14;14(2):139. doi: 10.3390/toxins14020139. PMID 35202166